CLINICAL TRIAL: NCT01351688
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD3514 in Japanese Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: An Open Label Prostate Cancer Study in Japanese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3760C00003
Record Dates: First submitted 2011-04-11; First posted 2011-05-11 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: Phase 1; Metastatic; Castration resistant; Prostate cancer; Androgen receptor; Down regulation; Japanese
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Bulbo-Spinal Atrophy, X-Linked | interventions — AZD3514

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD3514 (Experimental): Ascending doses of AZD3514 administered orally to patients to define the maximum tolerated dose (MTD)
  Interventions: Drug: AZD3514

INTERVENTIONS:
Drug: AZD3514 — Patients will be given AZD3514 tablets or capsules administered orally as a single dose, and then multiple once-daily dosing following a 7 day washout.

SUMMARY:
The primary aim of study is to gain an initial assessment of safety and tolerability of AZD3514 in Japanese patients together with assessing Pharmacokinetics (PK) and gaining a preliminary assessment of anti-tumour action. In this study, AZD3514 will be administered to Japanese patients with metastatic castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 20 years or older.
* Histologically or Cytologically proven diagnosis of prostate cancer for which no standard therapy is currently considered appropriate
* Documented evidence of metastatic prostate cancer
* Serum testosterone concentration ≤50 ng/dL
* World Health Organisation (WHO) performance status 0 to 1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks

Exclusion Criteria:

* History of hypersensitivity to active or inactive excipients of AZD3514 or drugs with a similar chemical structure or class to AZD3514
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD3514
* Inadequate bone marrow reserve or organ function
* Concurrent or recent treatment with certain medications or medical procedures
* Any medically important factors identified from electrocardiogram (ECG) measurements

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD3514 when given orally to Japanese patients with castration resistant prostate cancer | All AEs will be collected throughout the study, from informed consent until 30 days after the end of study treatment. The total duration of this time frame can not be specified
  Number of participants with adverse events

SECONDARY OUTCOMES:
To define the maximum tolerated dose, if possible, a lower biologically-effective dose(s) or maximum feasible dose of AZD3514 | during the single dose period and the first 21 days of multiple dosing (ie, by study day 29)
  A DLT is defined as any toxicity not attributable to the disease or disease-related processes under investigation and considered to be related to AZD3514 therapy during the single dose period and the first 21 days of multiple dosing (ie, by study day 29)
To characterise the pharmacokinetics of AZD3514 after a single oral dose and at steady state after multiple oral doses | Multiple timepoints taken, begining at Day 1 and until 48 hrs after last dose. The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
  To characterise the pharmacokinetics of AZD3514 after a single oral dose and at steady state after multiple oral doses
  * Cmax
  * Cmax at steady state (Cmax, ss)
  * time to maximum concentration (tmax)
  * tmax at steady state (tmax, ss)
  * terminal elimination rate constant (λz)
  * (AUC(0-t))
  * total clearance and terminal phase (Vz) of AZD3514
To obtain an preliminary assessment of the anti-tumour activity of AZD3514 | Every 12 weeks
To obtain an assessment of the activity of AZD3514 on the circulating levels of prostate-specific antigen (PSA) | Day 8, 15, 29 and every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glen Clack, MD, Study Director — AstraZeneca; Takefumi Sato, MD, Principal Investigator — Kitasato University
Locations (2):
- Japan (2):
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Sunto-gun, Shizuoka